CLINICAL TRIAL: NCT03184701
Title: Remote Monitoring of Symptoms and Cognitive Function Using Telehealth
Brief Title: Monitoring of Symptoms and Cognitive Function Using Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Victor Navarro, Chairman, Hepatology, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HN4828
Record Dates: First submitted 2017-03-30; First posted 2017-06-14 (Actual); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: End Stage Liver Disease
Keywords: Telehealth; Quality of Life
MeSH Terms: conditions — End Stage Liver Disease | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Patients assigned to this arm receive the intervention in addition to routine standard of care. Telehealth based remote monitoring of symptoms and brain tests is the intervention in this study. A device with preloaded questionaires will be given to patients randomized to this group. The patients will respond on a daily basis for the 3 months of intervention phase.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — Patients will be given an ipad with preloaded app (secured questions assessing their symptoms and cognitive function in a systematic timely way). The responses will be delivered to the care providers instantly, which will trigger an algorithmic clinical approach.

SUMMARY:
End-Stage Liver Disease (ESLD) is one of the ten leading causes of death in US. It is marked by episodic acute exacerbations of the underlying liver disease which often leads to severe symptoms, poor quality of life, mental deterioration and repeated hospitalizations.

The overall purpose of this project is to introduce a telehealth based intervention (involving remote monitoring of symptoms and cognitive function initiated at the time of discharge of ESLD patients. This will support enhanced clinical care and improve self-management in ESLD population. In addition, it will reduce healthcare utilization, improve medication adherence and overall health outcomes

DETAILED DESCRIPTION:
This is a single arm study to assess the effectiveness of an experimental telehealth intervention within the treatment of ESLD, and compare it with a historic cohort. All inpatients with advanced liver disease and at least 1 complication will be eligible to participate. the study group receives the Telehealth intervention and will be given an ipad preloaded with the instruments used for symptom monitoring and cognitive function assessment during the hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Liver Disease with at least 1 or more complications (Hepatorenal Syndrome, Portal Hypertension, Ascites, Hepatic Encephalopathy)

Exclusion Criteria:

* Cognitive impairment
* Current psychosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Navarro, MD, Principal Investigator — Einstein Healthcare network
Locations (1):
- Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: All study participants were included in this intervention arm, and given a device with questions to respond.
Period: Overall Study
Arm/Group | Intervention Arm
Started | 45
Completed | 28
Not Completed | 17
Not completed — Death | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: All participants are included in the study analyses.
Arm/Group | Experimental
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] | 55.7 [28 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 30
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Number of Participants reporting Satisfaction with Device
Time Frame: 3 months
Population: All participants who completed the end of study survey (at 3 months) are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 45
Participants | 45

2. Post Hoc Outcome: Hospital Readmissions at 30 Days
Description: Number of admissions to the hospital
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study participation (3 months)
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 3/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03184701/Prot_SAP_000.pdf